CLINICAL TRIAL: NCT06754605
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2 Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of Recombinant Respiratory Syncytial Virus Vaccine (SCTV02) in Healthy Adults ≥18 Years of Age
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Recombinant Respiratory Syncytial Virus Vaccine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCTV02-X201
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Syncytial Virus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- A: Low dose vaccine (Experimental): Low dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- A: Low dose placebo (Placebo Comparator): Placebo comparator of low dose, injected on Day 0
  Interventions: Biological: Placebo
- B: Medium dose vaccine (Experimental): Medium dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- B: Medium dose placebo (Placebo Comparator): Placebo comparator of medium dose, injected on Day 0
  Interventions: Biological: Placebo
- C: High dose vaccine (Experimental): High dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- C: High dose placebo (Placebo Comparator): Placebo comparator of high dose, injected on Day 0
  Interventions: Biological: Placebo
- D: Low dose vaccine (Experimental): Low dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- E: Medium dose vaccine (Experimental): Medium dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- F: High dose vaccine (Experimental): High dose of SCTV02, injected on Day 0
  Interventions: Biological: SCTV02
- G: Placebo (Placebo Comparator): Placebo comparator, injected on Day 0
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SCTV02 — Participants will receive a singe dose of SCTV02 on Day 0.
  Arms: A: Low dose vaccine; B: Medium dose vaccine; C: High dose vaccine; D: Low dose vaccine; E: Medium dose vaccine; F: High dose vaccine
Biological: Placebo — Participants will receive a singe dose of Placebo on Day 0.
  Arms: A: Low dose placebo; B: Medium dose placebo; C: High dose placebo; G: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled Phase 1/2 clinical trial to evaluate the safety, tolerability and immunogenicity of recombinant respiratory syncytial virus in participants aged 18 years and older.

DETAILED DESCRIPTION:
Three dose-levels of SCTV02 will be evaluated in participants aged 18 years and older. Solicited adverse events within 7 days post study vaccination and unsolicited adverse events within 30 days post study vaccination will be collected. Immunogenicity including Neutralizing antibody against RSV-A and RSV-B will be tested 14, 30, 90, 180 and 365 days post study vaccination will be assessed. T cell response will be tested 30 days post study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: male and female participants ≥18 years old at the time of signing the ICF; Phase II: male and female participants ≥50 years of age at the time of signing the ICF.
* Be able to sign a written Informed consent form (ICF) and participate in the trial voluntarily, and can fully understand the trial procedures and risks of participating in the trial.
* Be able to complete the diary card, contact card and diary/contact card by own or with the assistance of others.
* Phase I: healthy subjects or healthy subjects judged by the investigator according to the clinical data of the subjects; Stage II: Subjects who are healthy or have a stable underlying disease.
* Fertile men and women of childbearing age voluntarily agree to use effective contraception from the time they sign the ICF until 6 months after immunization; Pregnancy test results for women of childbearing age during the screening period were negative.

Exclusion Criteria:

* Acute illness and/or fever (axillary temperature ≥37.3 ° C) occurred within 3 days prior to vaccination with the study vaccine, or antipyretic, analgesic, or antiallergic drugs.
* Use any investigational or unregistered product within 30 days prior to immunization, or plan to use any such product during the study period.
* Concurrent participation in another clinical study where the subject has been or will be exposed to an investigational or non-investigational vaccine/product at any time during the study.
* Long-term or high-dose glucocorticoid therapy (duration ≥15 days, or dose ≥1 mg/kg/ day of prednisone or equivalent doses of other glucocorticoids), or other immunosuppressive and cytotoxic therapy within 90 days prior to vaccination.
* The study received a non-attenuated vaccine within 14 days prior to vaccination, or a live attenuated vaccine within 28 days; Have previously received the experimental respiratory syncytial virus (RSV) vaccine or been infected with RSV within 1 year prior to receiving the investigational vaccine.
* History or family history of epilepsy and mental illness.
* A family history of congenital or hereditary immunodeficiency, or a history and physical examination confirmed or suspected immunosuppression or immunodeficiency, or human immunodeficiency virus (HIV) infection, asplenia or functional asplenia.
* Have the following organ-specific or systemic autoimmune diseases: Guillain-Barre syndrome, myasthenia gravis, autoimmune hepatitis, ulcerative colitis, systemic lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome, and systemic sclerosis.
* Allergic to any component of the study vaccine, or any previous history of severe allergy to vaccine vaccination, such as anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, local allergic necrosis reaction, angioneurotic edema, etc.
* Severe chronic disease or active chronic disease, as assessed by the investigator, including but not limited to myocardial infarction, severe arrhythmia, unstable angina, uncontrolled blood pressure after medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg in subjects < 60 years of age; Hypertensive disease with systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg in subjects ≥60 years of age, diabetes mellitus with serious complications, cancer or precancerous lesions, and other serious cerebrovascular diseases, heart diseases, respiratory diseases, liver and kidney diseases, and thyroid diseases.
* Pregnant women (positive pregnancy test) or breastfeeding women, or those with pregnancy plans during the study period, or less than 6 weeks after the end of pregnancy (including ectopic pregnancy).

Plan to donate eggs or sperm during the study.

* Unable to follow the trial procedures, or plan to relocate or stay away for a long period of time during the study and cannot complete the trial follow-up.
* Any medical condition that makes intramuscular injection unsafe due to other abnormalities, conditions that may obfuscate the results of the study, or conditions that are not in the best interest of the subject, is determined by the investigator to be unsuitable for clinical study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of solicited adverse events within 7 days post study vaccination. | Day o to Day 7
  Incidence and severity of solicited adverse events within 7 days post study vaccination.
Geometric mean titer (GMT) of neutralizing antibodies (nAb) against RSV-A and RSV-B subtypes 30 days post vaccination | Day 30
  Geometric mean titer (GMT, Live Virus Neutralization Test) of neutralizing antibodies (nAb) against RSV-A and RSV-B subtypes 30 days after study vaccination.

SECONDARY OUTCOMES:
GMT of nAb against RSV-A and RSV-B subtypes 14 days after study vaccination.Immunogenicity 14 days post vaccination | Day 14
  GMT of nAb against RSV-A and RSV-B subtypes 14 days after study vaccination.
GMT of nAb against RSV-A and RSV-B subtypes 90 days post vaccination | Day 90
  GMT (Live Virus Neutralization Test) of neutralizing antibodies (nAb) against RSV-A and RSV-B subtypes 90 days after study vaccination.
GMT of nAb against RSV-A and RSV-B subtypes 180 days post vaccination | Day 180
  GMT (Live Virus Neutralization Test) of neutralizing antibodies (nAb) against RSV-A and RSV-B subtypes 180 days after study vaccination.
GMT of nAb against RSV-A and RSV-B subtypes 365 days post vaccination | Day 365
  GMT (Live Virus Neutralization Test) of neutralizing antibodies (nAb) against RSV-A and RSV-B subtypes 365 days after study vaccination.
T cell response | Day 30
  Number of T cell subsets activated by interferon-γ (for Th1) and interleukin-4 (for Th2) 30 days after study vaccination.
Incidence and severity of unsolicited adverse events within 30 days | Day to Day 30
  Incidence and severity of unsolicited adverse events within 30 days after study vaccination.
Incidence and severity of Serious adverse events and adverse events of special interest within 365 days | Day 0 to Day 365
  Incidence and severity of Serious adverse events and adverse events of special interest within 365 days after study vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Kexin, Doctor, Principal Investigator — Hebei Zhongshiyou Central Hospital
Locations (2):
- China (2):
  - Hebei Zhongshiyou Central Hospital, Langfang, Hebei
  - Luzhou Center for Disease Control and Prevention, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No